CLINICAL TRIAL: NCT00757744
Title: Behavioral Drug and HIV Risk Reduction Counseling in Methadone Patients in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Richard S. Schottenfeld, M.D., Yale University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0709003081; R01DA014718-05A1S1 (NIH)
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2011-05

CONDITIONS: Opiate Dependence; HIV Infections
Keywords: drug counseling; HIV risks; methadone maintenance; HIV Seronegativity
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Methadone maintenance treatment with Behavioral Drug and HIV Risk Reduction Counseling (BDRC)
  Interventions: Behavioral: Behavioral Drug and HIV Risk Reduction Counseling (BDRC)
- B (Active Comparator): Methadone maintenance treatment with standard drug counseling
  Interventions: Behavioral: Drug counseling

INTERVENTIONS:
Behavioral: Behavioral Drug and HIV Risk Reduction Counseling (BDRC) — once weekly individual counseling
  Arms: A
Behavioral: Drug counseling — individual drug counseling
  Arms: B

SUMMARY:
A randomized clinical trial evaluating the reduction of HIV risk behaviors and drug use when providing integrated behavioral drug and HIV risk reduction counseling (BDRC) along with methadone maintenance treatment in Wuhan, China

DETAILED DESCRIPTION:
This project is a supplement to a parent grant, Drug Counseling and Abstinence-Contingent Take-Home Buprenorphine in Malaysia. The specific aims of the parent grant include evaluating whether the relatively minimal counseling and other services provided with standard buprenorphine maintenance treatment (Standard BUP) is sufficient or whether one or a combination of two enhanced behavioral treatments--behavioral drug and HIV risk reduction counseling (BDRC) or abstinence-contingent take-home buprenorphine (ACB)-improve its efficacy (Specific Aim 1) and are cost-effective, with regard to the direct economic costs of providing the treatments (Specific Aim 2) and also to provide training and mentoring in drug abuse treatment and HIV prevention research to clinical researchers and clinical training for health professionals in Malaysia (Specific Aim 4). BDRC utilizes short-term behavioral contracts to promote abstinence and reduce drug- and sex-related HIV risk behaviors and can be provided by nurses and medical assistants available in medical settings in developing countries.

The specific aims of the proposed study are consistent with the specific aims of the parent grant and include evaluating in a pilot, randomized clinical trial in a methadone treatment program in Wuhan, China, the feasibility and potential efficacy for reducing illicit drug use and HIV risk behaviors of BDRC when combined with standard methadone treatment services (Standard Methadone) compared to Standard Methadone only (Specific Aim 1 of the proposed study). Additional Specific Aims of the proposed study include developing estimates of the treatment costs and cost-effectiveness of Standard Methadone and BDRC (Specific Aim 2 of the proposes study), and providing training and mentoring in drug abuse treatment and HIV prevention research to clinical researchers an clinical training for health professionals in China (Specific Aim 3 of the proposed study).

Specific aims of the China project:

1. Conduct a preliminary evaluation of the feasibility, acceptability, and preliminary efficacy for increasing treatment retention and reducing drug use and HIV risk behaviors of Behavioral Drug and HIV Risk Reduction Counseling (BDRC) when combined with Standard Methadone, in comparison to Standard Methadone, among opiate dependent treatment seeking volunteers admitted to the Wuhan Methadone Clinic.
2. Develop estimates of the costs and cost-effectiveness of Standard Methadone and BDRC.
3. Train and provide ongoing clinical supervision to a core group of 10 drug counseling staff and provide additional mentoring in drug abuse and HIV risk reduction research to investigators in China.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependence

Exclusion Criteria:

* current dependence on alcohol, benzodiazepines or sedatives
* current suicide or homicide risk
* current psychotic disorder or untreated major depression
* life-threatening or unstable medical problems

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Reductions of illicit opiate use | 6 months
Reductions in HIV risk behaviors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Schottenfeld, MD, Principal Investigator — Yale University
Locations (2):
- Yale University School of Medicine - CMHC, New Haven, Connecticut, United States
- Wuhan Center for Disease Control and Prevention, Wuhan, Hubei, China